CLINICAL TRIAL: NCT05664464
Title: A Phase Ib/II Randomized, Open Label Drug Repurposing Trial of Glutamate Signaling Inhibitors in Combination With Chemoradiotherapy in Patients With Newly Diagnosed Glioblastoma
Brief Title: Glutamate Inhibitors in Glioblastoma
Acronym: GLUGLIO
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-01877
Record Dates: First submitted 2022-12-07; First posted 2022-12-23 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Glioblastoma
Keywords: IDH wild-type; newly diagnosed; glutamate; epilepsy
MeSH Terms: conditions — Glioblastoma; Epilepsy | interventions — Gabapentin; Sulfasalazine; Memantine; Temozolomide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care (Active Comparator): Radiotherapy 30 x 2 Gy with concomitant temozolomide followed by maintenance temozolomide
  Interventions: Drug: Temozolomide; Radiation: Radiotherapy
- Standard of care plus glutamate signaling inhibitors (Experimental): Radiotherapy 30 x 2 Gy with concomitant temozolomide followed by maintenance temozolomide plus combined daily gabapentin, sulfasalazine and memantine
  Interventions: Drug: Gabapentin; Drug: Sulfasalazine; Drug: Memantine; Drug: Temozolomide; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Gabapentin — Weekly dose escalations over 4 weeks of daily 3 x 300 mg up to 3 x 1200 mg
  Arms: Standard of care plus glutamate signaling inhibitors
Drug: Sulfasalazine — Weekly dose escalations over 3 weeks of daily 3 x 500 mg up to 3 x 1500 mg
  Arms: Standard of care plus glutamate signaling inhibitors
Drug: Memantine — Weekly dose escalations over 4 weeks of daily 1 x 5-20 mg
  Arms: Standard of care plus glutamate signaling inhibitors
Drug: Temozolomide — Concomitant with radiotherapy at 75 mg/m2 daily followed by maintenance 150-200 mg/m2 on 5/28 days
Radiation: Radiotherapy — 30 x 2 Gy involved field radiotherapy with concomitant temozolomide

SUMMARY:
The goal of this 1:1 randomized, multi-center, open-label phase Ib/II clinical trial is to explore the efficacy of the add-on of the anti-glutamatergic drugs gabapentin, sulfasalazine and memantine to standard chemoradiotherapy with temozolomide compared to chemoradiotherapy alone in patients with newly diagnosed glioblastoma.

DETAILED DESCRIPTION:
Background: Glioblastoma is the most common and the most aggressive primary malignant brain tumor in adults. The clinical course of glioblastoma is invariably fatal despite multimodal therapy comprising surgical resection followed by chemoradiotherapy. Population-based median overall survival is in the range of only 12 months. Glioblastomas synthesize and secrete large quantities of the excitatory neurotransmitter glutamate, driving epilepsy, neuronal death, tumor growth and invasion.

Rationale: Several brain-penetrating drugs that have obtained clinical approval in other contexts can inhibit glutamate synthesis, secretion and signalling, including (i) the anti-epileptic drug gabapentin, which is a potent inhibitor of the critical glutamate synthesis enzyme branched chain amino acid transaminase 1 (BCAT-1), (ii) the anti-inflammatory drug sulfasalazine, which is a potent inhibitor of glutamate secretion by blocking the cystine-glutamate exchanger system Xc, and (iii) the cognitive enhancer memantine, which can prevent glutamate-driven, calcium-induced neuronal death and tumor cell invasion by blocking N-methyl-D-aspartate (NMDA) type glutamate receptors. The omnipresence and pleiotropic functions of glutamate in glioblastoma lends rationale for a combined anti-glutamatergic therapeutic approach. The well-documented tolerability of these drugs support the feasibility of a repurposing approach in combination with standard chemoradiotherapy. There is limited commercial interest in exploring the activity of these drugs as anti-cancer agents.

Aim: The aim of the herein proposed clinical trial is to explore the tolerability and efficacy of combined anti-glutamatergic treatment as an add-on to standard chemoradiotherapy in newly diagnosed glioblastoma. The trial is designed to explore the efficacy of a triple anti-glutamatergic treatment regimen to justify and statistically plan a subsequent phase III expansion trial.

Methodology: This randomized phase Ib/II, parallel-group, open-label, multicenter trial will be conducted in 120 adult patients with newly diagnosed glioblastoma. Any study treatments will be administered orally in combination with standard chemoradiotherapy and will be continued until tumor progression. The trial design comprises a per-patient dose-escalation approach in the experimental arm, i.e. doses of the study drugs will be increased weekly to pre-specified maximum dose levels and will be reduced if toxicities attributed to either study drug occur. The primary endpoint is progression-free survival at 6 months (PFS-6) and will be analysed by intent-to-treat. After the first 20 events in the experimental study arm, an interim toxicity analysis will be performed to evaluate study discontinuation and maximum target dose level adaptions. Secondary endpoints include estimates of median PFS and overall survival (OS), OS at 12 months, seizure-free survival (SFS) and SFS-6. Secondary objectives include the central review of neuropathological diagnoses, central response assessment on magnetic resonance imaging scans (MRI) utilizing the Response Assessment in Neuro-Oncology (RANO) working group criteria, determination of quality of life of patients and their care givers, symptom burden, cognitive functioning, anti-epileptic drug use, steroid use and exploratory analyses of outcome among molecular glioblastoma subtypes determined by methylome and gene panel sequencing.

ELIGIBILITY:
Inclusion criteria

* Diagnosis: Newly diagnosed supratentorial glioblastoma according to the 2021 World Health Organization (WHO) Classification of Central Nervous System Tumors
* Signed informed consent
* Age >18 years
* Eligible for standard chemoradiotherapy with temozolomide (TMZ/RT->TMZ, hypofractionated RT regimen not allowed)
* KPS 70 or more
* Ability to judge per local investigator estimate (at least oriented to time, place and situation)
* Paraffin-embedded tissue for central pathology review
* Adequate heamatological, liver and renal function

Exclusion criteria

* Scheduled for hypofractionated radiotherapy
* Women who are pregnant or breast feeding,
* Intention to become pregnant during the course of the study or intention to father a child,
* Lack of safe contraception, defined as: Female participants of childbearing potential, not using and not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the investigator in individual cases. Female participants who are surgically sterilised / hysterectomised or post-menopausal for longer than 2 years are not considered as being of child bearing potential.
* Other clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease),
* Known or suspected non-compliance, drug or alcohol abuse,
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* Participation in another study with investigational drug within the 30 days preceding and during the present study,
* Previous enrolment into the current study,
* Being an investigator, his/her family members, employees and other dependent persons,
* Any prior radiotherapy of the brain or radiotherapy with potential overlap of the irradiation fields,
* Active malignancy that may interfere with the study treatment,
* Abnormal ECG with QTc >450 ms,
* Contraindication for Gadolinium-enhanced MRI,
* Previous intolerance reactions to one of the study drugs,
* Intolerance reactions to sulfonamides or salicylates,
* Acute intermittend porphyria,
* Known glucose-6-phosphate dehydrogenase deficiency,
* Concomitant therapy with digoxin, cyclosporin, methotrexate,
* History of exfoliative dermatitis, Stevens-Johnson-Syndrome, toxic epidermal necrolysis, DRESS (Drug Rash with Eosinophilia and Systemic Symptoms) syndrome or renal tubular acidosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
PFS-6 | 6 months
  progression-free survival at 6 months

SECONDARY OUTCOMES:
PFS | From date of randomization until the date of first documented tumor progression or date of death from any cause, whichever came first, assessed for a minimum of 6 months and up to 42 months
  progression-free survival
OS | From date of randomization until the date of death from any cause, assessed for at least 6 months and up to 42 months
  overall survival
OS-12 | 12 months
  overall survival at 12 months
SFS | From date of randomization until the date of first documented seizure or date of death from any cause, whichever came first, assessed for a minimum of 6 months and up to 42 months
  Seizure-free survival
SFS-6 | 6 months
  Seizure-free survival at 6 months
QoL | From date of randomization until the date of first documented tumor progression or date of death from any cause, whichever came first, assessed for a minimum of 6 months and up to 42 months
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30 and Brain Tumor Module BN20 (EORTC QLQ-C30/BN20)
Symptom burden | From date of randomization until the date of first documented tumor progression or date of death from any cause, whichever came first, assessed for a minimum of 6 months and up to 42 months
  MD Anderson Symptom Inventory Brain Tumor (MDASI-BT) questionnaire, Neurologic assessment in neuro-oncology (NANO) scale
Quality of life of an informal caregiver | From date of randomization until the date of first documented tumor progression or date of death from any cause, whichever came first, assessed for a minimum of 6 months and up to 42 months
  CareGiver Oncology Quality of Life (CarGO-QOL) questionnaire
Cognitive Functioning | From date of randomization until the date of first documented tumor progression or date of death from any cause, whichever came first, assessed for a minimum of 6 months and up to 42 months
  Montreal Cognitive Assessment (MoCA) test

OTHER OUTCOMES:
Overall response rate | From date of randomization until the date of first documented tumor progression or date of death from any cause, whichever came first, assessed for a minimum of 6 months and up to 42 months
  as defined by RANO
Tumor glutamate levels | From date of randomization until the date of first documented tumor progression or date of death from any cause, whichever came first, assessed for a minimum of 6 months and up to 42 months
  determined by MRI spectroscopy
General condition | From date of randomization until the date of first documented tumor progression or date of death from any cause, whichever came first, assessed for a minimum of 6 months and up to 42 months
  Karnofsky Performance Status (KPS)
Anticonvulsant drug use and steroid use | From date of randomization until the date of first documented tumor progression or date of death from any cause, whichever came first, assessed for a minimum of 6 months and up to 42 months
  Documentation of drug name, dose, frequency and duration of intake
Subgroup survival analyses | From date of randomization until the date of first documented tumor progression, or death from any cause, whatever occurs first, assessed for at least 6 months and up to 42 months
  PFS compared between subgroups segregated by baseline parameters including age, extent of resection, KPS, MGMT promotor methylation status, steroid intake, presence or absence of seizures, tumor volumes, glutamate levels determined by MR spectroscopy, and molecular subtypes
Subgroup survival analyses | From date of randomization until the date of death from any cause, assessed for at least 6 months and up to 42 months
  OS compared between subgroups segregated by baseline parameters including age, extent of resection, KPS, MGMT promotor methylation status, steroid intake, presence or absence of seizures, tumor volumes, glutamate levels determined by MR spectroscopy, and molecular subtypes

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Georg Wirsching, MD, Principal Investigator — University Hospital and University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mastall M, Roth P, Bink A, Fischer Maranta A, Laubli H, Hottinger AF, Hundsberger T, Migliorini D, Ochsenbein A, Seystahl K, Imbach L, Hortobagyi T, Held L, Weller M, Wirsching HG. A phase Ib/II randomized, open-label drug repurposing trial of glutamate signaling inhibitors in combination with chemoradiotherapy in patients with newly diagnosed glioblastoma: the GLUGLIO trial protocol. BMC Cancer. 2024 Jan 15;24(1):82. doi: 10.1186/s12885-023-11797-z. PMID 38225589
- See also: Related Info — https://bmccancer.biomedcentral.com/articles/10.1186/s12885-023-11797-z